CLINICAL TRIAL: NCT04781452
Title: Evaluating the Treatment in the the Center for Disabled People in Aachen (MZEB Aachen) - a Registry on Patients With Severe Disabilities
Brief Title: Evaluating the Treatment in the MZEB Aachen
Acronym: EvalMZEB
Status: Recruiting | Type: Observational
Sponsor: RWTH Aachen University (Other)
Responsible Party: Principal Investigator, Andrea Maier, Principal Investigator, RWTH Aachen University
Other Study IDs: 19-006
Record Dates: First submitted 2020-01-09; First posted 2021-03-04 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Intellectual Disability; Disability Physical
MeSH Terms: conditions — Intellectual Disability

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: standard treatment — there ist no Intervention but our standart Treatment in the center

SUMMARY:
Evaluation of patient characteristics, involved physicians and therapists as well as therapies in a German University Center for the Treatment of patients with intellectual disabilities and severe multiple disability (MZEB Aachen)

DETAILED DESCRIPTION:
In the MZEB Aachen, since 11/2018 patients with intellectual disabilities and/or severe multiple disabilities are diagnosed, treated and accompanied for many years in a multidisciplinary setting with physicians, nurses, physiotherapists, ergo therapists, speech therapists and Support by social workers. MZEBs are considered to have a pilot function in the health care system, cooperating with therapists and physicians in the surroundings. This concept is established as a new concept in Germany in order to optimise health care for patients with disabilities. Thus we want to investigate patient characteristics, diagnoses, involved physicians and therapists as well as proposed therapies and disease progress in this center.

ELIGIBILITY:
Inclusion Criteria:

* intellectual disability and/or severe multiple disability (disability degree GdB at least 70 and at least one noticeable sign
* willing to participate

Exclusion Criteria:

* housed in an Institution and/or prison

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Mixed Population of People with intellectual and severe multiple disability who need this care in this center
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2029-07-01 (Estimated); Study Completion 2029-07-01 (Estimated)

PRIMARY OUTCOMES:
change in number of therapy sessions | baseline and after one year treatment
  change in the number of therapy sessions per month
Change in diagnoses | baseline and after one year treatment
  Change in percentage of definite diagnoses

CONTACTS AND LOCATIONS:
Overall Officials: Jörg B Schulz, MD, Study Chair — RWTH Aachen University
Locations (1):
- RWTH Aachen University, Aachen, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: Undecided
All relevant results will be shared

REFERENCES:
- See also: Web Address of the institution — http://www.mzeb.ukaachen.de